CLINICAL TRIAL: NCT06976450
Title: Evaluating the Effectiveness of ChemoNurs: A Mobile Chemotherapy Drug Guide for Oncology Nurses - A Randomized Controlled Trial
Brief Title: Evaluating the Effectiveness of ChemoNurs: A Mobile Chemotherapy Drug Guide for Oncology Nurses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Koç University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Enes Simsek, Principal Investigator, Koç University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2022.216.IRB3.099
Record Dates: First submitted 2025-05-09; First posted 2025-05-16 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-05

CONDITIONS: Chemotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: An independent statistician and a doctoral student working as a research assistant were responsible for the randomization and group assignment processes. Their involvement ensured the systematic conduct of the study and helped control selection bias through randomized allocation and allocation concealment. Due to the researcher's awareness of the intervention, blinding during the implementation phase was not feasible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Application Group (Experimental): Participants in the experimental group were oncology nurses employed at Hacettepe University Oncology Hospital who were provided access to CHEMONURS, a mobile chemotherapy drug guide application developed to support clinical decision-making and professional development. After completing a demographic form and baseline assessments using the Chemotherapy Practice Knowledge Scale and the Attitude Scale for Chemotherapy Practices, participants received a demo version of the app via a WhatsApp link. They were instructed to download the application onto their personal smartphones and use it freely over a six-month period during their routine clinical practice. No restrictions were placed on usage frequency to reflect real-world applicability; usage was monitored through embedded app analytics and nurse feedback. Daily reminders and follow-up communications were used to encourage continued engagement. Follow-up assessments of knowledge and attitudes were conducted at the 3rd and 6th months.
  Interventions: Other: ChemoNurs Mobile Application Group; Device: Personal Smartphone
- Standard Practice (No Intervention): Participants in the control group were oncology nurses working at Hacettepe University Oncology Hospital who continued with their routine clinical duties without access to the CHEMONURS mobile application or any additional educational intervention. After completing the baseline assessment using the Chemotherapy Practice Knowledge Scale and the Attitude Scale for Chemotherapy Practices, no further intervention was provided. Follow-up assessments of knowledge and attitudes were conducted at the 3rd and 6th months, in parallel with the experimental group, to evaluate changes over time in the absence of the mobile application.

INTERVENTIONS:
Other: ChemoNurs Mobile Application Group — Participants in the mobile app group were oncology nurses employed at Hacettepe University Oncology Hospital who were provided access to CHEMONURS, a mobile chemotherapy drug guide application developed to support clinical decision-making and professional development. After completing a demographic form and baseline assessments using the Chemotherapy Practice Knowledge Scale and the Attitude Scale for Chemotherapy Practices, participants received a demo version of the app via a WhatsApp link. They were instructed to download the application onto their personal smartphones and use it freely over a six-month period during their routine clinical practice. No restrictions were placed on usage frequency to reflect real-world applicability; usage was monitored through embedded app analytics and nurse feedback. Daily reminders and follow-up communications were used to encourage continued engagement. Follow-up assessments of knowledge and attitudes were conducted at the 3rd and 6th months. U
  Arms: Application Group
Device: Personal Smartphone — Used by participants to access and interact with the CHEMONURS mobile application during the study period.
  Arms: Application Group

SUMMARY:
This study aimed to evaluate the effectiveness of a mobile chemotherapy drug guide application, ChemoNurs, developed for oncology nurses, in improving their knowledge and attitudes toward chemotherapy practices.

H1: The mobile chemotherapy drug guide developed for oncology nurses increases their knowledge related to chemotherapy.

H2: The mobile chemotherapy drug guide developed for oncology nurses promotes the development of positive attitudes toward chemotherapy.

H3: The mobile chemotherapy drug guide developed for oncology nurses increases their satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Actively administering chemotherapy treatments
* Having knowledge of how to use an Android or iOS smartphone
* Possessing mobile literacy
* Working in oncology clinics for a duration of 0-12 months
* Volunteering to participate in the study

Exclusion Criteria:

* Not having completed the orientation process in oncology clinics
* Not having administered chemotherapy
* Incomplete responses in the data collection forms
* Willingness to withdraw at any stage of the study
* Participation in the Oncology Nursing Certification Program
* Prior attendance in courses or training sessions related to chemotherapy drugs

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Change in Chemotherapy Knowledge Score | Baseline (Month 0), Midpoint (Month 3), and Endpoint (Month 6)
  This outcome evaluates the improvement in oncology nurses' knowledge of chemotherapy administration, assessed through the Chemotherapy Practice Knowledge Scale for Oncology Nurses. The items are scored to assess nurses' knowledge related to chemotherapy practices using a 3-point Likert scale: "I have knowledge = 3," "I am unsure = 2," and "I have no knowledge = 1." The scale consists of 44 items and four subdimensions. The total score ranges from a minimum of 44 to a maximum of 132, with higher scores indicating greater knowledge regarding chemotherapy administration.
Change in Attitudes Toward Chemotherapy Practices | Baseline (Month 0), Midpoint (Month 3), and Endpoint (Month 6)
  This outcome measures changes in the attitudes of oncology nurses toward chemotherapy practices, using the Attitude Scale for Oncology Nurses Regarding Chemotherapy Practices. This scale was developed by Khan et al. (2012) to evaluate the attitudes of cancer nurses toward chemotherapy practices. It is a 4-point Likert-type scale with the following response options: 4 = Strongly Agree, 3 = Agree, 2 = Disagree, 1 = Strongly Disagree. The scale consists of two subdimensions: negative attitude (6 items) and positive attitude (4 items). The items under the negative attitude subdimension are reverse-scored when calculating the total score. The overall score ranges from a minimum of 10 to a maximum of 40, with higher scores indicating more positive attitudes toward chemotherapy practices.

SECONDARY OUTCOMES:
Mobile Application Usability | Month 3 and Month 6
  Evaluation of the usability of the CHEMONURS mobile application as assessed by the Mobile Application Usability Scale at Month 3 and Month 6. The scale was created by Hoehle et al. (2016), and its Turkish adaptation was made by Güler in 2019. This tool provides information about the colors, text styles, font sizes, transitivity, application management, etc., used in the mobile application. The scale is a 7-point Likert-type measurement tool and consists of a total of 40 questions. The minimum score is 40, and the maximum score is 280, with higher scores indicating better usability.
Nurses' Satisfaction with CHEMONURS Application | Month 6
  Nurses' overall satisfaction with the CHEMONURS mobile application, assessed using the Satisfaction Scale at the end of the study (Month 6). To evaluate cancer nurses' satisfaction with the ChemoNurs mobile application, they were asked at the end of the sixth month to rate their satisfaction on a scale from 1 to 10, where 1 = Not at all satisfied and 10 = Very satisfied. Higher scores indicate better satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Remziye Semerci Şahin, Assistant professor, Study Director — Koç University
Locations (1):
- Hacettepe University Oncology Hospital, Ankara, Altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No